CLINICAL TRIAL: NCT04145466
Title: The Personalized Nutrition Study: Evaluation of a Genetically-informed Weight Loss Approach
Brief Title: The Personalized Nutrition Study
Acronym: POINTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Principal Investigator, Corby K. Martin, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBRC 2019-043
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Diet, High-Fat; Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel arm trial with 4 groups over 12 weeks
  1. Fat responders receiving a high-fat diet (n=52)
  2. Fat responders receiving a high-carbohydrate diet (n=52)
  3. Carbohydrate responders receiving a high-fat diet (n=25)
  4. Carbohydrate responders receiving a high-carbohydrate diet (n=25)
  The total number per group is an estimate. We will not close cells to enroll this exact number per group, and the total number of people enrolled will not exceed 154.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to diet assignment and genotype pattern. Interventionists will be blind to genotype pattern, but not diet type. To enhance external validity, participants will be told if they are carbohydrate or fat responders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fat responders (1) (Experimental): receiving high-fat diet
  Interventions: Behavioral: High-fat diet
- Carbohydrate responders (1) (Experimental): receiving high-fat diet
  Interventions: Behavioral: High-fat diet
- Fat responders (2) (Experimental): receiving high-carbohydrate diet
  Interventions: Behavioral: High-carbohydrate diet
- Carbohydrate responders (2) (Experimental): receiving high-carbohydrate diet
  Interventions: Behavioral: High-carbohydrate diet

INTERVENTIONS:
Behavioral: High-fat diet — The high-fat diet will consist of ~40% energy from fat and ~45% from carbohydrates. Protein will be 15% of energy.
  All participants will be assigned an energy intake target that will result in a daily deficit of ~750 kcal, though no energy intake targets below 1,100 kcal/d (women) and 1,300 kcal/day (men) will be prescribed
  Arms: Carbohydrate responders (1); Fat responders (1)
Behavioral: High-carbohydrate diet — The high-carbohydrate diet will consist of ~20% of energy from fat and ~65% from carbohydrates. Protein will be 15% of energy.
  All participants will be assigned an energy intake target that will result in a daily deficit of ~750 kcal, though no energy intake targets below 1,100 kcal/d (women) and 1,300 kcal/day (men) will be prescribed
  Arms: Carbohydrate responders (2); Fat responders (2)

SUMMARY:
A person's genetic code is believed to affect how much weight he/she will lose during diets that vary in carbohydrate and dietary fat content. 'Carbohydrate responders' are hypothesized to lose more weight on diets that are high in carbohydrates, as compared to high in fats. 'Fat responders' are hypothesized to lose more weight on diets that are high in dietary fat, as compared to high in carbohydrates. The purpose of the proposed study is to test these hypotheses in a randomized controlled trial.

DETAILED DESCRIPTION:
Obesity and its comorbidities are major public health challenges. To combat the obesity pandemic, many weight-loss strategies have been studied, often emphasizing either high carbohydrate (low fat) diets or high fat (low carbohydrate) diets. Mean weight loss differences between high-carbohydrate and high-fat diets that induce equal caloric deficits have been reported to be small; however, the individual weight loss response varies substantially within diet groups, suggesting that different individuals react differently to high-carbohydrate or high-fat diets. This assumption is supported by retrospective data showing that participants with carbohydrate-responsive polymorphisms lost 2-3 times more weight when assigned to a high-carbohydrate diet compared to a high-fat diet, and vice versa for those with dietary fat-responsive polymorphisms. Conversely, a recent randomized clinical trial aimed to determine the effect of a healthy high-fat diet (high in unsaturated fats) vs. a healthy high-carbohydrate diet (high in whole-grain foods) on 12-month weight change but did not find significant differences between the two groups and failed to find the hypothesized association between genotype patterns and weight loss induced by diets that varied in fat and carbohydrate content. However, an important caveat of their approach is that the single nucleotide polymorphisms selected by the investigators had not been previously associated with obesity or with dietary responses, which may explain their lack of predictive value in identifying differences in inter-individual responses. In addition, the fat composition of the diets was relatively high in both high- and low-fat groups. The inconsistent findings in the literature indicate a need for further research to determine if genetic factors affect weight loss when exposed to diets that vary in carbohydrates and dietary fats.

The purpose of this randomized controlled parallel arm trial is to test the following hypotheses.

Hypothesis 1 will test if participants assigned to the diet that corresponds to their genotype lose more weight than those assigned to a diet inconsistent with their genotype.

Hypothesis 2 will analyze the fat responders and carbohydrate responders separately.

* Hypothesis 2a: Fat responders will lose more weight on the high-fat diet vs. the high-carbohydrate diet.
* Hypothesis 2b: Carbohydrate responders will lose more weight on the high-carbohydrate diet vs. the high-fat diet.

Carbohydrate responders and fat responders will be randomized to one of the following two diets:

1. A high-quality high-carbohydrate diet that is rich in whole-grain foods, or
2. A high-quality high-fat diet that is rich in unsaturated fats and oils

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27.0 kg/m2 to < 47.5 kg/m2
* Completed genealogy test and access to the raw data
* Fat responder or Carbohydrate responder, as determined by genetic risk score

It is estimated that approximately 1/3 of people are fat responders, 1/3 are carbohydrate responders, and 1/3 are neither or will respond to either diet. Only carbohydrate and fat responders are eligible.

Exclusion Criteria:

* Current smoker or has smoked in the previous year
* For females, pregnant or planned pregnancy during the study duration, or breast-feeding, based on self-report
* Conditions, diseases, or medications that affect body weight or metabolism (e.g., certain antipsychotic medications; type 2 diabetes mellitus; heart failure; cancer, excluding certain melanomas; etc.)
* Has gained or lost more than 10 pounds in the last 3 months
* Currently diagnosed with an eating disorder, major depression, or other condition that, in the judgment of the investigators, could affect the risk to the participant or study completion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Access to individual de-identified data is possible via Pennington Biomedical Research Center's Data Sharing policy.

REFERENCES:
- [Derived] Hochsmann C, Yang S, Ordovas JM, Dorling JL, Champagne CM, Apolzan JW, Greenway FL, Cardel MI, Foster GD, Martin CK. The Personalized Nutrition Study (POINTS): evaluation of a genetically informed weight loss approach, a Randomized Clinical Trial. Nat Commun. 2023 Oct 9;14(1):6321. doi: 10.1038/s41467-023-41969-1. PMID 37813841

RESULTS

PARTICIPANT FLOW:
Groups:
- Fat Responders (1); Carbohydrate Responders (1): receiving high-fat diet
  High-fat diet: The high-fat diet will consist of ~40% energy from fat and ~45% from carbohydrates. Protein will be 15% of energy.
  All participants will be assigned an energy intake target that will result in a daily deficit of ~750 kcal, though no energy intake targets below 1,100 kcal/d (women) and 1,300 kcal/day (men) will be prescribed
- Fat Responders (2); Carbohydrate Responders (2): receiving high-carbohydrate diet
  High-carbohydrate diet: The high-carbohydrate diet will consist of ~20% of energy from fat and ~65% from carbohydrates. Protein will be 15% of energy.
  All participants will be assigned an energy intake target that will result in a daily deficit of ~750 kcal, though no energy intake targets below 1,100 kcal/d (women) and 1,300 kcal/day (men) will be prescribed
Period: Overall Study
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2)
Started | 50 | 23 | 49 | 23
Completed | 46 | 22 | 43 | 18
Not Completed | 4 | 1 | 6 | 5

BASELINE CHARACTERISTICS:
Population: Includes participants that completed the study and were included in the analysis. Of the 129 participants that completed the study, 7 participants were incorrectly genotyped and were not included in the final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2) | Total
Number analyzed (Participants) | 44 | 21 | 41 | 16 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.5) | 49.8 (14.1) | 54.4 (14.2) | 52.4 (13.0) | 54.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 17 | 35 | 13 | 102
  Male | 7 | 4 | 6 | 3 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 9 | 10 | 5 | 36
  White | 30 | 12 | 31 | 10 | 83
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 3
Weight [Mean (Standard Deviation); unit: kg] | 94.2 (14.0) | 95.2 (17.6) | 93.5 (14.4) | 95.6 (18.1) | 94.3 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Weight (kg) at 12 weeks minus weight at baseline (kg)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2)
Number analyzed (Participants) | 44 | 21 | 41 | 16
kg | -5.5 (1.2) | -4.1 (1.7) | -5.3 (1.3) | -5.1 (1.6)

2. Primary Outcome: Percent Weight Change
Description: Weight change (kg) / weight at baseline (kg) * 100
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2)
Number analyzed (Participants) | 44 | 21 | 41 | 16
percent | -5.9 (1.3) | -4.8 (1.9) | -5.7 (1.4) | -5.7 (1.8)

3. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference (cm) at 12 weeks minus waist circumference at baseline (cm)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2)
Number analyzed (Participants) | 44 | 21 | 41 | 16
cm | -5.0 (1.4) | -4.2 (2.3) | -4.4 (1.5) | -4.4 (2.1)

4. Secondary Outcome: Change in Food Cravings
Description: Food cravings are assessed via the total score of the 33-item Food Craving Inventory (FCI). The FCI is scaled in a frequency format, assessing the frequency with which an individual experiences a craving for a particular food. All items are scored in the following manner: Never = 1, Rarely = 2, Sometimes = 3, Often = 4, & Always = 5. Responses from all 33 items are then averaged to produce a total score (range 1-5). Lower total scores indicate a low frequency of cravings across several food groups including high fat foods, sweets, carbohydrates, fast food fats, and fruits and vegetables while higher total scores indicate a high frequency of cravings across these food groups.
  Change in food cravings is calculated as FCI total score at 12 weeks minus FCI total score at baseline.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2)
Number analyzed (Participants) | 41 | 19 | 38 | 13
score on a scale | -0.3 (0.2) | -0.5 (0.2) | -0.3 (0.2) | 0.0 (0.2)

5. Secondary Outcome: Change in Fat Preference Index
Description: Preference for high- versus low-fat foods is measured with the 74-item Food Preference Questionnaire (FPQ). Individual items in the FPQ measure the preference for either a high fat food or a low fat food on a 9-point Likert scale with the following anchors: 1 = dislike extremely; 5 = neutral, neither like nor dislike; 9 = like extremely.
  The fat preference index (range: 1/9 - 9) is then calculated as the mean rating for high-fat foods divided by the mean rating for low-fat foods. Values greater than 1.0 reflect a higher fat preference, and values less than 1.0 reflect a lower fat preference.
  Change in Fat Preference Index is calculated as Fat Preference Index at 12 weeks minus Fat Preference Index at baseline.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2)
Number analyzed (Participants) | 44 | 21 | 41 | 16
score on a scale | 0.0 (0.4) | 0.0 (0.5) | 0.0 (0.5) | -0.2 (0.5)

6. Secondary Outcome: Change in Disinhibition
Description: Score on the Disinhibition subscale (16-items) of the 36-item Three-Factor Eating Questionnaire. Items are scored as 'true'=1 or 'false'=0. The Disinhibition score (range: 1-16) is calculated as a sum score of all items within that subscale such that low scores indicate more inhibition while higher scores indicate more disinhibition
  Change in Disinhibition is calculated as the score on the Disinhibition subscale at 12 weeks minus the score on the Disinhibition subscale at baseline.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2)
Number analyzed (Participants) | 37 | 18 | 31 | 12
score on a scale | -0.3 (0.8) | 0.0 (0.9) | 0.2 (0.9) | 0.7 (0.9)

7. Secondary Outcome: Change in Hunger
Description: Score on the Hunger subscale (14 items) of the 36-item Three-Factor Eating Questionnaire. Items are scored as 'true'=1 or 'false'=0. The Hunger score (range: 1-14) is calculated as a sum score of all items within that subscale such that low scores indicate a lower tendency to be hungry while higher scores indicate a greater tendency to be hungry.
  Change in Hunger is calculated as the score on the Hunger subscale at 12 weeks minus the score on the Hunger subscale at baseline.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2)
Number analyzed (Participants) | 37 | 18 | 31 | 14
score on a scale | -0.9 (0.7) | -0.1 (0.9) | -1.3 (0.8) | 0.8 (0.8)

8. Secondary Outcome: Change in Cognitive Restraint
Description: Score on the Cognitive Restraint subscale (21 items) of the 36-item Three-Factor Eating Questionnaire. Items are scored as 'true'=1 or 'false'=0. The Cognitive Restraint score (range: 1-21) is calculated as a sum score of all items within that subscale such that low scores indicate less cognitive restraint while higher scores indicate greater cognitive restraint.
  Change in Cognitive Restraint is calculated as the score on the Cognitive Restraint subscale at 12 weeks minus the score on the Cognitive Restraint subscale at baseline
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2)
Number analyzed (Participants) | 34 | 18 | 29 | 12
score on a scale | 3.5 (1.2) | 4.6 (1.1) | 2.7 (1.4) | 3.4 (1.1)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Fat Responders (1) | Carbohydrate Responders (1) | Fat Responders (2) | Carbohydrate Responders (2)
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/22 | 0/43 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/46 | 0/22 | 1/43 | 0/18
Other Adverse Events (participants affected / at risk) | 0/46 | 0/22 | 2/43 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fat Responders (1) (N=46) | Carbohydrate Responders (1) (N=22) | Fat Responders (2) (N=43) | Carbohydrate Responders (2) (N=18)
Hospitalized (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Admitted to hospital 3/18/2021 to drain abscess on colon. History of diverticulitis. D/C'd on 03/21/2021 and back home.
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Diagnosed with RSV and was hospitalized due to difficulty breathing.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fat Responders (1) (N=46) | Carbohydrate Responders (1) (N=22) | Fat Responders (2) (N=43) | Carbohydrate Responders (2) (N=18)
Lymphodema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Lymphodema diagnosed after a surgery to repair a broken leg. The surgery was in Dec. 2020.
Lipedema (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Lipedema and fluid retention. Prior ankle surgery cause of this (before POINTS participation). Weight fluctuating frequently.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT04145466/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT04145466/ICF_001.pdf